CLINICAL TRIAL: NCT07226297
Title: An Open-label Single Center, Single Participant Study of an Experimental Antisense Oligonucleotide Treatment for Charcot-Marie-Tooth Type 2D Due to GARS1 Genetic Mutation
Brief Title: Personalized Antisense Oligonucleotide for A Single Participant With GARS1 Gene Mutation Associated With Charcot-Marie-Tooth Disease Type 2D (CMT2D)
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-25-0625
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Charcot-Marie-Tooth Disease Type 2D
MeSH Terms: conditions — Charcot-Marie-Tooth disease, Type 2D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: nL-GARS1-001

INTERVENTIONS:
Drug: nL-GARS1-001 — Personalized antisense oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single participant with Charcot-Marie-Tooth disease type 2D (CMT2D) due to a pathogenic, de novo deletion mutation in GARS1

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single participant with CMT2D due to a pathogenic, de novo deletion mutation in GARS1

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or the participant's parent(s) or legally authorized representative(s).
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records.

Genetically confirmed GARS1 genetic variant

Exclusion Criteria:

* Participant has any condition that, in the opinion of the Site Investigator, would ultimately prevent the completion of study procedures.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Motor Skills | Baseline to 24 months
  Change in fine motor skills from baseline to 12- and 24-months post nL-GARS1-001 administration as measured by the annualized rate of change in the Nine-Hole Peg Test (9-HPT)
Motor Skills | Baseline to 24 months
  Change in fine motor skills from baseline to 12- and 24-months post nL-GARS1-001 administration as measured by the annualized rate of change in the Box and Block Test (BBT)
Motor Skills | Baseline to 24 months
  Change in gross motor skills from baseline to 12- and 24-months post nL-GARS1-001 administration as measured by the annualized rate of change on Revised Upper Limb Module (RULM)
Motor Skills | Baseline to 24 months
  Change in gross motor skills from baseline to 12- and 24-months post nL-GARS1-001 administration as measured by the annualized rate of change on Hammersmith Functional Motor Scale - Expanded (HFMSE)
Motor Skills | Baseline to 24 months
  Change in gross motor skills from baseline to 12- and 24-months post nL-GARS1-001 administration as measured by the annualized rate of change on home videography assessment

SECONDARY OUTCOMES:
Quality of Life | Baseline to 24 months
  Change in quality of life from baseline to 6-, 12-, 18- and 24-months post nL-GARS1-001 administration as measured by the Pediatric Quality of Life Inventory (PedsQL)
Functional Skills | Baseline to 24 months
  Change in functional skills from baseline to 6-, 12-, 18- and 24-months post nL-GARS1-001 administration as measured by the Pediatric Evaluation of Disability Inventory - Computer Adaptive Test (PEDI-CAT)
Safety and Tolerability | Baseline to 24 months
  Incidence and severity of treatment-emergent adverse events (AEs) post nL-GARS1-001 administration
Incidence of Treatment-Emergent Abnormalities in Physical Exam [Safety and Tolerability] | Baseline to 24 months
  Changes post nL-GARS1-001 administration in physical examination (changes in appearance, skin, neck, ears, nose, throat, heart/lungs, abdomen, lymph nodes, and extremities compared to baseline)
Incidence of Treatment-Emergent Abnormalities in Neurological Exam [Safety and Tolerability] | Baseline to 24 months
  Changes post nL-GARS1-001 administration in neurological examination (changes in mental status, gait, cerebellar, cranial nerve, motor, reflex, and sensations compared to baseline as assessed by treating physician)
Incidence of Treatment-Emergent Abnormalities in Safety Labs (CSF, chemistry, hematology, coagulation, and urinalysis) [Safety and Tolerability] | Baseline to 24 months
  Emergent abnormalities in laboratory analyses (results outside of normal range for CSF, chemistry, hematology, coagulation, and urinalysis)

OTHER OUTCOMES:
Pulmonary Function | Baseline to 24 months
  Change in Forced Vital Capacity (FVC) from baseline to 12- and 24-months post nL-GARS1-001 administration
Pulmonary Function | Baseline to 24 months
  Change in Forced Expiratory Volume in 1 second (FEV1) from baseline to 12- and 24-months post nL-GARS1-001 administration
Nerve Function | Baseline to 24 months
  Change in nerve function from baseline to 12- and 24-months post nL-GARS1-001 administration as measured by speed and strength of electrical signals in the motor and sensory nerves
Cognition | Baseline to 24 months
  Change in cognition from baseline to 12- and 24-months post nL-GARS1-001 administration as measured by NIH Toolbox Cognition assessment
Communication | Baseline to 24 months
  Change in communication skills from baseline to 12- and 24-months post nL-GARS1-001 administration as measured by the Communication Participation Item Bank (CPIB)

CONTACTS AND LOCATIONS:
Locations (1):
- UTHealth Houston, Houston, Texas, United States